CLINICAL TRIAL: NCT05036122
Title: Validation of a Non-Invasive Instrument to Estimate Blood Lactate
Brief Title: Estimating Blood [Lactate] Non-Invasively
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-000318
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: High intensity exercise; Stress Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Whole-body exercise in healthy adults (Aim 1) (Experimental): Subjects will have blood [lactate] measurement obtained with the LabClasp device while completing an exercise stress test on a treadmill or bicycle.
  Interventions: Device: LabClasp
- ICU patients susceptible to developing sepsis (Aim 2) (Experimental): Subjects will have blood [lactate] measurement obtained with the LabClasp device as frequently as required for clinical purposes
  Interventions: Device: LabClasp

INTERVENTIONS:
Device: LabClasp — Non-invasive device that estimates blood [lactate] from interstitial fluid via a proprietary algorithm. The device is placed between the first and second knuckle of a finger and gently applies slight pressure to extract interstitial fluid from the skin. Sensors within the device quickly estimate blood [lactate] and return a value to the subject via an accompanying tablet within 20 seconds.

SUMMARY:
The purpose of this study is to validate the LabClasp's ability to estimate blood [lactate].

ELIGIBILITY:
Inclusion Criteria - Aim 1:

* Subjects must be able to provide written consent.
* Adults 18 years of age and older.
* Nonsmokers.
* No recent hospitalization (< 60 days).
* Ability to perform high-intensity exercise.

Inclusion Criteria - Aim 2:

* Subjects must be able to provide written consent to be included in the research study.
* Adults 18 years of age and older.
* Nonsmokers.
* Current ICU patient.
* Have regular blood samples taken for [lactate] measurements.
* Have one or more risk factors for sepsis.

Exclusion Criteria - Aims 1 and 2:

* History of, or active malignancy.
* History of HIV with antiretroviral treatment.
* Smokers.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood [lactate] during incremental exercise | 1 day
  Measured via venous blood and the LabClasp
Blood [lactate] measurements in ICU patients | 1 day
  Measured via venous blood and the LabClasp

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States